CLINICAL TRIAL: NCT03941054
Title: Treatment of Myosfascial Trigger-Points of Gastrocnemius and Its Effects on the Neuromuscular Response
Brief Title: Myosfascial Trigger-Points and Effects on Neuromuscular Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Albert Pérez Bellmunt, Director, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Protocol ID : P3/03
Record Dates: First submitted 2019-05-03; First posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Myofascial Trigger Point Pain
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): No intervention
- Pressure Release (Experimental): Digitopressure treatment of the Myosfascial Trigger Points
  Interventions: Other: Pressure Release

INTERVENTIONS:
Other: Pressure Release — Subjets receive digitopressure during 90 seconds for the treatment of the Myosfascial Trigger Points
  Arms: Pressure Release

SUMMARY:
The aim of this study is to analyze the effects of the treatment of the Myosfascial Trigger-Points detected in the gastrocnemius muscles on the neuromuscular response.

ELIGIBILITY:
Inclusion Criteria:

* Subjets with both active or latent Myosfascial Trigger Points

Exclusion Criteria:

* Pregnant women
* Musculoskeletal problems in the last month
* Surgical interventions in he knee, hip, ankle, back or neck in tha last 6 months
* Psychological or nervous alterations
* Uncomprehension of the study protocol

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2019-06-07 (Estimated); Study Completion 2019-06-07 (Estimated)

PRIMARY OUTCOMES:
change of neuromuscular stiffness of the gastrocnemious muscles | 10 minutes before the intervention, and 1 minute after the intervention
  biomechanical property of a muscle that characterizes the resistance to an external force that deforms its initial shape, using a "Myoton".
change of elasticity of the gastrocnemious muscles | 10 minutes before the intervention, and 1 minute after the intervention
  Biomechanical property of a muscle that characterizes the ability to recover its initial shape after the removal of the external force that lead to its deformation, using a "Myoton".
change of relaxation of the gastrocnemious muscles | 10 minutes before the intervention, and 1 minute after the intervention
  Time for a muscle to recover its shape from deformation after the removal of an external force, using a "Myoton".

SECONDARY OUTCOMES:
change of active dorsiflexion ROM | 4 minutes before the intervention, and 6 minute after the intervention
  Active range of movement of the dorsiflexion of the ankle, using an inclinometer (degrees).
change of pasive dorsiflexion ROM | 2 minutes before the intervention, and 8 minute after the intervention
  Pasive range of movement of the dorsiflexion of the ankle, using an inclinometer (degrees).
change of gastrocnemious strength | 5 minutes before the intervention, and 5 minute after the intervention
  Isometric strength of the gastrocnemious muscles using a handheld dynamometer "microFET 2" (newtons).
change of pain intensity | 8 minutes before the intervention, and 2 minute after the intervention
  How much pressure needs to be applied to cause pain
change of pressure-pain threshold | 7 minutes before the intervention, and 3 minute after the intervention
  How much pain the pacient reports while a pressure of 1kg/cm²/s is being applied over his gastrocnemious muscle

CONTACTS AND LOCATIONS:
Overall Officials: Albert Pérez-Bellmunt, PhD, Principal Investigator — Anatomy lecturer
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No